CLINICAL TRIAL: NCT02345135
Title: Susceptibility to Infections in Patients With Ataxia Telangiectasia : A Prospective Follow-up Study
Brief Title: Susceptibility to Infections in Ataxia Telangiectasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Stefan Zielen, Prof. Dr. med., Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INFECTION_AT2012
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Ataxia Telangiectasia; Infections; Immunodeficiency; Lung Disease
MeSH Terms: conditions — Ataxia Telangiectasia; Infections; Immunologic Deficiency Syndromes; Lung Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ataxia Telangiectasia (Active Comparator): All A-T patients presented for 3 study visits. In all visits patients had a clinical examination, a blood collection and a lung function measurement. Furthermore symptom diaries were distributed and collected on these visits.
  Interventions: Procedure: Blood collection; Procedure: Lung function measurement; Behavioral: Symptom diary
- Healthy Control (Active Comparator): All healthy controls presented for 3 study visits. In all visits patients had a clinical examination and a lung function measurement. Furthermore symptom diaries were distributed and collected on these visits.
  Interventions: Procedure: Lung function measurement; Behavioral: Symptom diary

INTERVENTIONS:
Procedure: Blood collection — In all patients with Ataxia telangiectasia blood was collected at each visit date to determine blood count, lymphocyte subpopulation count and immunoglobulin levels in serum (IgA, IgG, IgM, IgE), as well as alpha feto protein (AFP).
  Arms: Ataxia Telangiectasia
Procedure: Lung function measurement — In all patients - Ataxia telangiectasia and healthy controls - a lung function measurement was done to determine vital capacity (VC), forced expiratory volume in 1 second (FEV1), peak expiratory flow (PEF) and Tiffenau index.
Behavioral: Symptom diary — All patients - Ataxia telangiectasia and healthy controls - were requested to keep a symptom diary for the months September to March of the years 2012/2013 and 2013/2014 to determine days with symptoms as coughing during day and night, cold and fever, as well missing days at kindergarten/school/work, intake of medication (especially antibiotic treatment) and hospitalisations.

SUMMARY:
Death in Ataxia telangiectasia (A-T) is usually due to cancer or chronic lung failure around 20 years of age. Despite low lymphocyte counts (CD3, CD4, CD8 and CD19), IgA and IgG subclass deficiency opportunistic and acute severe respiratory infections are rare. The prevailing wisdom is that an immunoglobulin replacement therapy is not necessary in most of the patients. However no placebo controlled trials have been performed so far. The aim of this trial was to investigate the prevalence of mild and severe respiratory infections and / or chronic cough in classical A-T patients compared to healthy controls.

DETAILED DESCRIPTION:
Ataxia telangiectasia is an autosomal recessive multisystem disorder which is characterized by a progressive ataxia, conjunctival telangiectasia, a humoral and cellular immunodeficiency, an increased radiosensitivity and an increased risk for cancer (Boder E, Pediatrics, 1957). Most patients die in their 2nd or 3rd decade of life due to a respiratory failure caused by progressive (interstitial) lung disease or due to malignancies (Schroeder SA, Pediatr Pulmonol, 2010). In 1995 the sequence of the mutated AT gene (ATM) on chromosome 11q22-23 was identified. Main problems besides the progressive neurodegeneration are recurrent infections of upper and lower respiratory tract and a growth retardation and malnutrition. These problems are caused by a mutation in the ATM gene on chromosome 11, which encodes for a protein with several key functions in control of cell cycle and apoptosis (Savitsky K et al., Hum Mol Gen, 1995). Several works already showed that patients with AT have a variable immunodeficiency which is characterized by low lymphocyte counts, a lack of Immunoglobulin A (IgA), Immunoglobulin G subclasses (IgG2 and 4) and specific pneumococcal antibodies (Schubert R, Clin Exp Immunol, 2002). The course of disease is dependent on the AT mutation respectively the residual kinase activity of ATM which is found in about 10% of A-T patients. These patients are described as 'variant ATs´ and have a better prognosis regarding immunodeficiency, susceptibility to infections and a possible growth retardation and malnutrition (Verhagen M, Hum Mutat, 2012). Despite the evidence for a humoral immunodeficiency a treatment with polyvalent immunoglobulins (IgG) is not practiced in generally. In the 'Clinical Workshop on Ataxia Teleangiectasia´, that took place in Frankfurt in January 2011, the investigators found out that the percentage of A-T patient, that are supplemented with immunoglobulins was only 10% to 60% depending on the different clinical centres.The Goethe University Childrens Hospital in Frankfurt, the biggest A-T centre in Germany, takes care for more than 40 A-T patients. At the moment about 15% of these patients are treated with immunoglobulins. Some observations show that the progress of the chronic lung disease cannot be prevented the usage of immunoglobulins. By now it´s not clear in what way patients suffer from an increased susceptibility to infections and if a substitution with immunoglobulins is needed. The aim of this trial is to investigate the incidence, intensity and duration of infections in patients with A-T compared to age matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* A-T: clinically and/or genetically diagnosed A-T
* No IgG treatment from the point of being included into the study
* Healthy controls: healthy children or adults matched for gender and age
* age 2 - 45 years
* written informed consent

Exclusion Criteria:

* age < 2 or > 45 years
* patient has to be treated with IgG-replacement regularly
* Other diseases with influence on the immune system (e.g. diabetes mellitus, malignancy, dialysis-dependent renal failure)

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2012-09; Primary Completion 2016-01-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Number of days with a symptom score > 3 compared to healthy subjects matched for age. | 24 months

SECONDARY OUTCOMES:
Number of days of absence in kindergarten, school or at work | 24 months
Number of cold periods | 24 months
Number of antibiotic therapies | 24 months
Number of severe infections | 24 months
  Number of severe infections defined as abscess-forming pneumonia/meningitis and/or other infection with need for hospitalization compared to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof. Dr., Principal Investigator — Johann Wolfgang Goethe University, Childrens Hospital

REFERENCES:
- [Background] Schroeder SA, Zielen S. Infections of the respiratory system in patients with ataxia-telangiectasia. Pediatr Pulmonol. 2014 Apr;49(4):389-99. doi: 10.1002/ppul.22817. Epub 2013 Jun 13. PMID 23761391
- [Background] Schubert R, Reichenbach J, Rose M, Zielen S. Immunogenicity of the seven valent pneumococcal conjugate vaccine in patients with ataxia-telangiectasia. Pediatr Infect Dis J. 2004 Mar;23(3):269-70. doi: 10.1097/01.inf.0000115737.35353.55. PMID 15014308
- [Background] McGrath-Morrow SA, Gower WA, Rothblum-Oviatt C, Brody AS, Langston C, Fan LL, Lefton-Greif MA, Crawford TO, Troche M, Sandlund JT, Auwaerter PG, Easley B, Loughlin GM, Carroll JL, Lederman HM. Evaluation and management of pulmonary disease in ataxia-telangiectasia. Pediatr Pulmonol. 2010 Sep;45(9):847-59. doi: 10.1002/ppul.21277. PMID 20583220
- [Background] Schroeder SA, Swift M, Sandoval C, Langston C. Interstitial lung disease in patients with ataxia-telangiectasia. Pediatr Pulmonol. 2005 Jun;39(6):537-43. doi: 10.1002/ppul.20209. PMID 15789441
- [Background] Driessen GJ, Ijspeert H, Weemaes CM, Haraldsson A, Trip M, Warris A, van der Flier M, Wulffraat N, Verhagen MM, Taylor MA, van Zelm MC, van Dongen JJ, van Deuren M, van der Burg M. Antibody deficiency in patients with ataxia telangiectasia is caused by disturbed B- and T-cell homeostasis and reduced immune repertoire diversity. J Allergy Clin Immunol. 2013 May;131(5):1367-75.e9. doi: 10.1016/j.jaci.2013.01.053. Epub 2013 Apr 6. PMID 23566627
- [Background] Verhagen MM, Martin JJ, van Deuren M, Ceuterick-de Groote C, Weemaes CM, Kremer BH, Taylor MA, Willemsen MA, Lammens M. Neuropathology in classical and variant ataxia-telangiectasia. Neuropathology. 2012 Jun;32(3):234-44. doi: 10.1111/j.1440-1789.2011.01263.x. Epub 2011 Oct 24. PMID 22017321
- [Derived] Zielen S, Duecker RP, Woelke S, Donath H, Bakhtiar S, Buecker A, Kreyenberg H, Huenecke S, Bader P, Mahlaoui N, Ehl S, El-Helou SM, Pietrucha B, Plebani A, van der Flier M, van Aerde K, Kilic SS, Reda SM, Kostyuchenko L, McDermott E, Galal N, Pignata C, Perez JLS, Laws HJ, Niehues T, Kutukculer N, Seidel MG, Marques L, Ciznar P, Edgar JDM, Soler-Palacin P, von Bernuth H, Krueger R, Meyts I, Baumann U, Kanariou M, Grimbacher B, Hauck F, Graf D, Granado LIG, Prader S, Reisli I, Slatter M, Rodriguez-Gallego C, Arkwright PD, Bethune C, Deripapa E, Sharapova SO, Lehmberg K, Davies EG, Schuetz C, Kindle G, Schubert R. Simple Measurement of IgA Predicts Immunity and Mortality in Ataxia-Telangiectasia. J Clin Immunol. 2021 Nov;41(8):1878-1892. doi: 10.1007/s10875-021-01090-8. Epub 2021 Sep 3. PMID 34477998
- See also: German AT-website — http://www.info-at.de